CLINICAL TRIAL: NCT02227849
Title: An Open-Label, Multicenter Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of Canagliflozin (TA-7284) as add-on to GLP-1 Analogue in Subjects With Type 2 Diabetes Mellitus
Brief Title: Long-Term Safety Study of Canagliflozin (TA-7284) in Combination With GLP-1 Analogue in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-7284-12
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin (TA-7284) ＋GLP-1 analogue (Experimental)
  Interventions: Drug: Canagliflozin (TA-7284); Drug: GLP-1 analogue

INTERVENTIONS:
Drug: Canagliflozin (TA-7284) — The patients will receive Canagliflozin orally for 52 weeks
Drug: GLP-1 analogue

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Canagliflozin (TA-7284) in combination with GLP-1 analogue in patients with type 2 Diabetes for 52 weeks.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the long-term safety and efficacy of Canagliflozin (TA-7284) in Japanese patients with type 2 diabetes mellitus, who are receiving treatment with GLP-1 analogue on diet and exercise and have inadequate glycemic control. The patients will receive TA-7284 100mg orally for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been receiving a stable dose and regimen of GLP-1 analogue over 12 weeks before administration of investigational dug
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients with HbA1c of ≥7.0% and <10.5%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug

Exclusion Criteria:

* Patients with type 1 diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (Cushing's syndrome, acromegaly, etc.)
* Patients with severe diabetic complications (proliferative diabetic retinopathy, stage 4 nephropathy, or serious diabetic neuropathy)
* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg
* Patients with serious renal or hepatic disease
* Patients with eGFR of <45 mL/min/1.73 m2
* Patients who are the excessive alcohol addicts
* Patients requiring insulin therapy
* Patients who are pregnant, lactating and probably pregnant patients and patients who can not agree to contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuya Inagaki, Professor, Study Director — Kyoto University, Graduate School of Medicine; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (4):
- Japan (4):
  - Reserch site, Chūbu
  - Reserch site, Hokkaido
  - Reserch site, Kanto
  - Reserch site, Kinki

REFERENCES:
- [Result] Harashima SI, Inagaki N, Kondo K, Maruyama N, Otsuka M, Kawaguchi Y, Watanabe Y. Efficacy and safety of canagliflozin as add-on therapy to a glucagon-like peptide-1 receptor agonist in Japanese patients with type 2 diabetes mellitus: A 52-week, open-label, phase IV study. Diabetes Obes Metab. 2018 Jul;20(7):1770-1775. doi: 10.1111/dom.13267. Epub 2018 Mar 24. PMID 29473709

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin (TA-7284) + GLP-1 Analogue: Canagliflozin (TA-7284) 100mg once daily for 52 weeks in combination with GLP-1 analogue
Period: Overall Study
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Started | 71
Completed | 63
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessed by Adverse Events (Number of Participants Experiencing With Adverse Events)
Time Frame: 52 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 71
Participants
  Serious Adverse Event | 5
  Adverse Event | 51

2. Secondary Outcome: Change in Percentage of HbA1c
Time Frame: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 71
percentage of HbA1c | -0.70 (0.82)

3. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward. Outcome measure for one patient was not assessed at a certain timepoint due to dropout.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 70
mg/dL | -34.7 (37.7)

4. Secondary Outcome: Percentage Change in Body Weight
Time Frame: Baseline, 52 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 70
percent change | -4.46 (3.20)

5. Secondary Outcome: Change in Blood Pressure
Time Frame: Baseline, 52 Weeks
Population: Full analysis set, last observation carried forward.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Number analyzed (Participants) | 71
mmHg
  Systolic blood pressure | -7.90 (11.83)
  Diastolic blood pressure | -4.32 (8.00)

ADVERSE EVENTS:
Arm/Group | Canagliflozin (TA-7284) + GLP-1 Analogue
Serious Adverse Events (participants affected / at risk) | 5/71
Other Adverse Events (participants affected / at risk) | 43/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin (TA-7284) + GLP-1 Analogue (N=71)
Erysipelas (Infections and infestations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin (TA-7284) + GLP-1 Analogue (N=71)
Gastroenteritis (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 24
Pharyngitis (Infections and infestations) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pollakiuria (Renal and urinary disorders) | 6
Polyuria (Renal and urinary disorders) | 4
Contusion (Injury, poisoning and procedural complications) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other